CLINICAL TRIAL: NCT00863213
Title: Study of Ablation Versus antiaRrhythmic Drugs in Persistent Atrial Fibrillation
Acronym: SARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Medtronic (Industry); Fundacio Clinic Barcelona (Other); Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, MD Phd, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARA-08; EudraCT: 2008-006095-30
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation, Radiofrequency; Atrial fibrillation; Antiarrhythmic Drugs
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atrial Fibrillation Ablation (Experimental)
  Interventions: Procedure: Atrial fibrillation ablation
- Drug therapy (Active Comparator)
  Interventions: Drug: Antiarrhythmic drug

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Atrial fibrillation ablation with radiofrequency, guided by 3D navigation map. Either 4mm or cooled tip-catheters will be used.
  It will include, at least, pulmonary veins isolation; all other radiofrequency lines, including roof and mitral isthmus line, and complex fractioned electrograms ablation will be performed according to each Hospital protocol. Radiofrequency lines block will be tested.
  Arms: Atrial Fibrillation Ablation
Drug: Antiarrhythmic drug — Usual drug therapy for atrial fibrillation. In patients with structural heart disease, amiodarone is recommended, while flecainide plus diltiazem or beta-blockers are encouraged in patients without structural heart diseases.
  Arms: Drug therapy

SUMMARY:
The purpose of this study is to compare the effectivity and safety of atrial fibrillation ablation, in comparison to antiarrhythmic drug therapy in patients with refractory, persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent atrial fibrillation (more than 7 days, or less than 7 days needing pharmacologic or electric cardioversion)

Exclusion Criteria:

* Hypo or hyperthyroidism
* Persistent atrial fibrillation lasting more than 1 year or non-defined duration
* Hypertrophic myocardiopathy
* Implantable defibrillation or pacemaker implanted
* Moderate or severe mitral valve disease or mitral prosthetic valve
* Ejection fraction less than 30%
* Left atrial anteroposterior diameter more than 50 mm.
* Previous atrial fibrillation ablation
* Contraindication to anticoagulation
* Left atrium thrombus
* Current infective disease or sepsis
* Pregnant women
* Current unstable angor
* Acute myocardial infarction in last 3 months
* Atrial fibrillation secondary to ionic disturbance, thyroids disease or secondary to any other reversible or non cardiovascular disease
* Reduced expectancy of life (less than 12 months)
* Patient participating in another clinical study that investigates a drug or device
* Psychologically unstable patient or denies to give informed consent
* Any cause that contraindicate ablation procedure or antiarrhythmic drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmias, lasting more than 24 hours or requiring cardioversion. | 1-year follow-up

SECONDARY OUTCOMES:
Freedom from atrial arrhythmias (lasting more than 30 seconds) without antiarrhythmic drugs. | 1-year follow-up
Decrease in frequency and duration of atrial fibrillation or atrial flutter recurrences. | 1-year follow-up
Decrease in atrial fibrillation/atrial flutter related hospital admissions | 1-year follow-up
Improve in quality of life measured with standard questionary for Atrial Fibrillation: AF-QoL. | 1-year follow-up
Change in need of cardioversions | From 3rd to 12th months
Need of atrio-ventricular node ablation | 1-year follow-up
Need of crossover to the other arm of the study (only when primary end point has been reached) | 1-year follow-up
Need of a new intervention or ablation during blanking period | Until 3rd month
Detection of asymptomatic episodes by Reveal XT | 1-year follow-up
Presence of any complications in the acute phase or during follow-up | 1-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Mont, MD, Study Chair — Hospital Clinic of Barcelona; Angel Arenal, MD, Study Director — Hospital Gregorio Marañon; Julian Villacastin, MD, Study Director — Hospital San Carlos, Madrid; Josep Brugada, prof Md. PHD, Study Director — Hospital Clinic of Barcelona
Locations (8):
- Spain (8):
  - Hospital Clinic Universitari, Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital de Cruces, Bilbao, Bizkaia
  - Clínica Puerta de Hierro, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid

REFERENCES:
- [Derived] Mont L, Bisbal F, Hernandez-Madrid A, Perez-Castellano N, Vinolas X, Arenal A, Arribas F, Fernandez-Lozano I, Bodegas A, Cobos A, Matia R, Perez-Villacastin J, Guerra JM, Avila P, Lopez-Gil M, Castro V, Arana JI, Brugada J; SARA investigators. Catheter ablation vs. antiarrhythmic drug treatment of persistent atrial fibrillation: a multicentre, randomized, controlled trial (SARA study). Eur Heart J. 2014 Feb;35(8):501-7. doi: 10.1093/eurheartj/eht457. Epub 2013 Oct 17. PMID 24135832